CLINICAL TRIAL: NCT06720233
Title: A Phase III, Multicenter, Open-label, Single-arm Clinical Study to Evaluate the Efficacy and Safety of SAL-0951 Tablets in the Treatment of Renal Anemia in Patients With Chronic Kidney Disease Receiving Maintenance Peritoneal Dialysis
Brief Title: Efficacy and Safety Study of SAL-0951 in the Treatment of Renal Anemia in Patients Receiving Peritoneal Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAL0951A303
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Anemia
Keywords: Anemia; Renal Insufficiency; Chronic Dialyses; Peritoneal Dialysis; Enarodustat
MeSH Terms: conditions — Anemia; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAL-0951 tablets (Experimental): initial phase：4mg QD subsequent phase：1mg～8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Interventions: Drug: SAL-0951 tablets

INTERVENTIONS:
Drug: SAL-0951 tablets — initial phase：4mg QD subsequent phase：1mg～8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Other Names: SAL-0951 group

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of SAL-0951 in Chinese patients receiving peritoneal dialysis with chronic kidney disease and anemia

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-arm clinical study (using individualized dose adjustment design). Eligible subjects after screening will be assigned to the test group for a 24-week treatment to verify the efficacy and safety of SAL-0951 in the treatment of renal anemia in patients receiving peritoneal dialysis.

The study is mainly divided into four stages: screening period (2 or 4 weeks before administration), initial treatment period (4 weeks), maintenance treatment period (20 weeks), and safety follow-up period (2 weeks), requiring a total of 11 visits. This study includes the 24th week visit as the end of treatment visit (EOT) and the 26th week as the end of study visit (EOS). Subjects who withdraw early will be required to complete the research procedure for Week 24.

ELIGIBILITY:
Inclusion Criteria:

1.Dry weight 45 to 100 kg; 2.Patients receiving continuous peritoneal dialysis for at least 12 weeks prior to the screening visit and no other blood purification treatment (including hemodialysis) within 12 weeks prior to the screening visit; 3.Patients continuing on peritoneal dialysis during the period between the screening visit and the end of study, without receiving other blood purification treatment (including hemodialysis); 4.Patients with TSAT*1 >20% or ferritin*1 >50 μg/L at screening visit;

* 1: Invalid test values cannot be used to determine a subject's eligibility. If serum iron values are invalid values, TSAT values shall also be handled as invalid values and re-test will be performed (For patients with ferritin >50 μg/L, there is no need for re-test).

  5.Patients who have received ESAs within 8 weeks prior to screening visit should meet the following requirements simultaneously* (* those with use of darbepoetin alfa (DA) prior to screening should meet all of the following 4 criteria, and those with use of rHuEPO prior to screening should meet both criteria #2 and #4):
  1. If the treatment drug is DA prior to the screening visit 1, the most recent treatment before the screening visit should be performed 2 weeks (including 2 weeks) prior to the screening visit 1;
  2. Treatment prescription regimen (including rHuEPO or DA, in which DA needs to be administered on the day of visit 1) consistent with the most recent ESAs prior to screening should be received at the screening visit 1 (same ESAs should be administered at the same dose; if the weekly dose is uneven in the regimen of the most recent ESAs prior to screening, for example, rHuEPO 5000 IU and 3000 IU are injected once every week alternately, proceed the treatment as per original regimen in the screening period; if rHuEPO is originally administered multiple doses weekly and the date of recent dose is less than 3 days from the day of the first dose of study drug, rHuEPO should be discontinued; if rHuEPO is originally administered weekly, the day of rHuEPO administration should be 3 days before the day of the first dose of study drug. Among them, rHuEPO of different brands is regarded as the same kind of ESAs. The acceptable average weekly dose is ≥750 IU and ≤9000 IU in a cycle of treatment based on the last prescription prior to screening, usually 4 weeks.);
  3. If the treatment drug is DA prior to screening visit 1, the acceptable average weekly dose is 10 µg to 30 µg in a cycle of treatment based on the last prescription of DA prior to screening, usually 4 weeks. It is not expected to receive DA from the day after screening visit 1 until the first dose of study drug according to the original dosing regimen, except in exceptional cases*1;
* 1: The same DA regimen adopted at screening visit 1 will be administered (at the same dose, using same drug) approximately 2 weeks after screening visit 1, provided that the time interval from the most recent DA therapy prior to screening visit 1 to screening visit 1 is less than 3 weeks (≥14 days and <21 days), and the screening period is 4 weeks.

  4)Patients with Hb levels ≥95 g/L and ≤120 g/L at the screening visit; 6.Patients not treated with ESAs (ESAs-naïve) within 12 weeks prior to the screening visit should meet the following a) and b) requirements:
  1. Patients not treated with ESAs during the period between screening visit 1 and the date of first dose of study drug
  2. Patients with Hb levels ≥80 g/L and ≤105 g/L at the screening visit 7.Voluntary participation in the trial and signature of informed consent.

Exclusion Criteria:

1. Patients with peritoneal dialysis catheter problems (dislocation, etc.), peritonitis, peritoneal dialysis catheter infection, etc. during the period between 4 weeks prior to the screening visit and the first dose of study drug, affecting the continuation of peritoneal dialysis;
2. Patients with poorly controlled hypertension (e.g., systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥110 mmHg at screening visit);
3. Patients with severe hepatobiliary disease (e.g., AST or ALT >2.5 × upper limit of normal value at screening visit, hepatic cirrhosis, total bilirubin ≥1.5 × upper limit of normal value at screening visit);
4. Patients with congestive heart failure (New York Heart Association [NYHA] Class III or greater) or unstable angina during the period between 24 weeks prior to the screening visit and the first dose of study drug;
5. Patients who have developed myocardial infarction, transient ischemic attacks, cerebral infarction (excluding asymptomatic cerebral infarction), or venous thromboembolism (pulmonary embolism or deep vein thrombosis) during the period between 24 weeks prior to the screening visit and the first dose of study drug;
6. Patients who will undergo an ophthalmological procedure (laser photocoagulation therapy or vitreous surgery) for the treatment of diabetic retinopathy, diabetic macular edema, or age-related macular degeneration during the period between screening visit and the end of the study;
7. Patients who have undergone erythrocyte transfusion during the period between 12 weeks prior to the screening visit and the first dose of study drug (as clinically indicated, transfusions of blood products that do not contain red blood cells may be excluded, such as plasma, albumin, etc.)
8. Subjects who have received growth hormone, thyroxine, testosterone enanthate, or mepitiostane during the period between 12 weeks prior to the screening visit and the first dose of study drug;
9. Patients with severe hyperparathyroidism (e.g., intact-parathyroid hormone [intact-PTH] ≥500 pg/mL at screening visit);
10. Patients with severe infections (such as active pulmonary tuberculosis, fungal infections, etc.), systemic hematological diseases (such as myelodysplastic syndrome, aplastic anemia, abnormal hemoglobin disease, etc.) or hemolytic anemia, or patients with anemia caused by bleeding disorders (such as gastrointestinal bleeding, etc.);
11. Except for glomerulonephritis, anemia patients suspected to be caused by non-infectious chronic inflammatory diseases such as systemic lupus erythematosus, rheumatoid arthritis, celiac disease, etc.;
12. Patients with polycystic kidney disease, any previous functional organ transplantation or scheduled organ transplantation;
13. Patients positive for any of the following: human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), or anti-hepatitis C virus antibodies (anti-HCV Ab), or confirmed syphilis requiring treatment;
14. Patients with medical history of malignancy (including hematological malignancy), except for tumors determined to be cured or in remission for 5 years, skin basal cell or squamous cell carcinoma that has undergone radical resection, or in situ carcinoma of any part;
15. Patients with a history of severe drug allergies (such as anaphylactic shock), or allergy to other HIF-PH inhibitors;
16. History of drug or alcohol abuse in the past two years*;

    *An average of 14 units of alcohol per week (1 unit ≈ 360 mL of beer, or 45 mL of liquor, or 150 mL of wine) in 2 years before screening
17. Patients who have received another investigational product (or study drug), have received treatment with an investigational device (or study device), or have participated in clinical research involving intervention (medical action beyond the scope of ordinary medical practice intended for research purposes) and received treatment during the period between 12 weeks prior to the screening visit and the first dose of study drug;
18. Patients who have received treatment with other HIF-PH inhibitors within 8 weeks prior to the screening or have previously participated in a clinical study of SAL-0951 and received the investigational product (active drug);
19. Patients who are pregnant, lactating, or may be pregnant (the possibility of pregnancy cannot be ruled out by the investigator based on the results of pregnancy test at screening visit);
20. Women of childbearing potential or men with sexual partners of childbearing potential who do not agree to take effective contraception* from the time of signing the informed consent until the end of the dosing study;

    *Effective contraceptive methods include transdermal patches, oral medication, implantable or injectable contraceptives, abstinence or birth control surgery.
21. Any other medical condition that, in the opinion of the investigator, could pose a safety risk to the subject in this study, could confound efficacy or safety assessment, or could interfere with the subject's participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2002-02-22 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Mean Hb level and 95% CI during the evaluation period after the 24-week treatment period or at the end of treatment | at Weeks 20, 22, and 24 [or end-of-treatment date]
  (Hb levels during the evaluation period are defined as the mean value of Hb levels at Weeks 20, 22, and 24 [or end-of-treatment date])

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, Ph.D, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No